CLINICAL TRIAL: NCT04865224
Title: Non-Invasive Estimation of Hemoglobin Levels in Blood Using Combined Deep Learning Methods
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Hakan Yılmaz, Asst. Prof. (Ph.D.), Karabuk University
Other Study IDs: B17EUni-2020-34
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Hemoglobin Level Measurement; Hemoglobin Level Estimation
Keywords: non-invasive; deep learning; hemoglobin level estimation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: hemoglobin estimation — In this method, in which different deep learning models are used together, the age range is intended to be as wide as possible to provide a quick solution with a high accuracy and low error values.

SUMMARY:
Hemoglobin is an important protein that gives the blood its red color and helps transport oxygen to organs. There are quite a lot of people in the world who need to have their hemoglobin levels checked regularly, especially anemia patients. It is important to keep the hemoglobin levels in the blood of these individuals under control. For this, it is necessary to measure in frequent periods. A large group, from adults to children, needs to take these measurements. Most of these are invasive measurements made with blood that require devices and trained people. These painful methods are quite uncomfortable.

In this study, non-invasive hemoglobin level measurement was aimed with a combined DL model created by using nail images with age, height, weight, BMI, and gender information of the volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Individuals need to be healthy.
* Individuals should not have any active hand or nail disease.
* Individuals should know their hemoglobin level.

Exclusion Criteria:

-In case of any condition that hides the natural nail color, such as henna, nail polish, protective or trauma-induced dents, bruises on the nails of individuals, it is removed from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People whose hemoglobin level has been measured in the clinic or laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Bland-Altman analysis | 1 day
  Bland-Altman analysis was performed to make the results simpler and more understandable. This analysis is especially used in the simple and graphical expression of measurements in which two methods are compared.
Estimation accuracy analysis | 1 day
  It is an analysis that compares the estimated hemoglobin values with the measured hemoglobin values.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No